CLINICAL TRIAL: NCT02288416
Title: Pilot Study of a Video-Based Intervention to Reduce Psychological Harm Associated With Lung Cancer Screening
Brief Title: Video-Based Intervention in Reducing Anxiety in Patients Undergoing Lung Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14169; NCI-2014-02220 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14169 (Other: City of Hope Medical Center)
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Anxiety; No Evidence of Disease; Lung Carcinoma
MeSH Terms: conditions — Anxiety Disorders; Lung Neoplasms | interventions — Early Intervention, Educational; Methods; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (standard of care) (Active Comparator): Patients receive standard of care following LCS consisting of routine visits and telephone contact with the LCS program nurse practitioner and coordinator.
  Interventions: Other: questionnaire administration; Other: quality-of-life assessment; Other: Best Practice
- Group II (video-based intervention) (Experimental): Patients undergo a video-based intervention prior to undergoing LCS. Patients watch a 5-minute video that focuses on preparing patients for LCS by providing information on the following: program team and contact information; reason to be screened; screening eligibility; how screening is performed; what to expect on the day of screening; what to expect after screening; what to expect if result is positive; what to expect if result is negative; and risks of screening. Patients also receive an educational handbook. Patients with positive scans (a Lung-RADS 3 or 4) receive additional brochure and nursing support within 1 week after notification of scan results.
  Interventions: Other: educational intervention; Other: questionnaire administration; Other: quality-of-life assessment

INTERVENTIONS:
Other: educational intervention — Undergo video-based intervention
  Other Names: intervention, educational
  Arms: Group II (video-based intervention)
Other: questionnaire administration — Ancillary studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: Best Practice
  Other Names: standard of care; standard therapy
  Arms: Group I (standard of care)

SUMMARY:
This pilot trial studies a video-based intervention in reducing anxiety in patients undergoing lung cancer screening. Giving a video-based intervention to patients prior to lung cancer screening may reduce anxiety and improve the well-being and quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the feasibility and acceptability of the video-based intervention.

SECONDARY OBJECTIVES:

I. To describe incidence, degree, and duration of screen-related anxiety among individuals scheduled to undergo low-dose computed tomography (CT) scan (LDCT) for lung cancer screening (LCS).

II. To describe baseline patient characteristics and pre-screening anxiety levels.

III. To describe the preliminary outcomes on screen-related anxiety for patients both not in the intervention group and those in the intervention group.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP I: Patients receive standard of care following LCS consisting of routine visits and telephone contact with the LCS program nurse practitioner and coordinator.

GROUP II: Patients undergo a video-based intervention prior to undergoing LCS. Patients watch a 5-minute video that focuses on preparing patients for LCS by providing information on the following: program team and contact information; reason to be screened; screening eligibility; how screening is performed; what to expect on the day of screening; what to expect after screening; what to expect if result is positive; what to expect if result is negative; and risks of screening. Patients also receive an educational handbook. Patients with positive scans (a Lung-Imaging Reporting and Data Systems [RADS] 3 or 4) receive additional brochure and nursing support within 1 week after notification of scan results.

After completion of LCS, patients are followed up at 1 week and then at 3 and 7 months.

ELIGIBILITY:
Inclusion Criteria:

* This study will be conducted in people scheduled to undergo baseline LDCT as part of the City of Hope (COH) LCS program
* There are no restrictions related to performance status and life expectancy
* All subjects must have the ability to understand and the willingness to participate in the informed consent process, although a waiver of written informed consent is obtained for this study

Exclusion Criteria:

* Patients who do not speak or read, because all intervention materials, including the video and written materials are in English
* Subjects, who in the opinion of the investigator, may not be able to comply with study procedures

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12-08; Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Percent of patients who complete the intervention | Baseline
  Descriptive statistics will be presented on participation in all components of the intervention.
Patient satisfaction with the timing, content, and delivery of the video-based intervention assessed by survey | Up to 7 months
  This self-reported measure will be completed by subjects who received the intervention.

SECONDARY OUTCOMES:
Patient screen-related anxiety as assessed by the mean score of the State Trait Anxiety Inventory (STAI) | Baseline to 7 months
  The survey is used to diagnose anxiety and to distinguish it from depressive syndromes, with items rated on a 4-point scale (with 1 being "Almost Never" and 4 being "Almost Always").
Health-related quality of life as assessed by the mean survey score of the Short Form-12 (SF-12) questionnaire | Up to 7 months
  The SF-12 is designed for assessment of general health status and contains 7 items that measure physical functioning, role functioning, bodily pain, energy/fatigue, social functioning, mental health, emotional functioning, general health perceptions, and changes in health.
Consequences of screening, assessed by the mean survey score of the Consequences of Screening in Lung Cancer (COS-LC) questionnaire | Up to 7 months
  This questionnaire is a non-validated adapted version of a validated two part tool used to assess the psychological impact to breast cancer screening using mammography.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Raz, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States